CLINICAL TRIAL: NCT02844816
Title: Phase II Trial of Atezolizumab in BCG-Unresponsive Non-Muscle Invasive Bladder Cancer
Brief Title: Atezolizumab in Treating Patients With Recurrent BCG-Unresponsive Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01104; NCI-2016-01104 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1605 (Other: SWOG); S1605 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Results first posted 2023-12-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Bladder Urothelial Carcinoma; Stage 0a Bladder Urothelial Carcinoma AJCC v6 and v7; Stage 0is Bladder Urothelial Carcinoma AJCC v6 and v7; Stage I Bladder Urothelial Carcinoma AJCC v6 and v7
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab) (Experimental): Patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles (51 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq

SUMMARY:
This phase II trial studies how well atezolizumab works in treating patients with non-muscle invasive bladder cancer that has come back (recurrent) and has not responded to treatment (refractory) with Bacillus Calmette-Guerin (BCG). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate complete response at 25 weeks after registration for those with a carcinoma in situ (CIS) component and to evaluate event-free survival at 18 months in patients with BCG-unresponsive high-risk non-muscle invasive bladder cancer (Ta/T1/CIS) treated with atezolizumab.

SECONDARY OBJECTIVES:

I. To estimate event-free survival at 18 months for the subset of patients with papillary cancer (Ta/T1).

II. To estimate progression-free survival, cystectomy-free survival, bladder cancer-specific survival, overall survival in all patients.

ADDITIONAL OBJECTIVES:

I. To estimate the level of agreement between local and central pathology review in terms of recurrence (for all patients) and complete response (for the CIS subset).

II. To identify markers that predict response to atezolizumab in the CIS population and that are associated with event-free survival (EFS) in patients with Ta/T1/CIS BCG-unresponsive non-muscle invasive bladder cancer. The following markers will be tested:

IIIa. Expression of PD-L1 and CD8 by immunohistochemistry (IHC). IIIb. Expression of immune signatures by ribonucleic acid (RNA)-sequencing (RNA-seq).

IIIc. Peripheral immune response by mass cytometry (CyTOF) and TruCulture.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles (51 weeks) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 2 years and then every 24 weeks for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven, recurrent, non-muscle invasive urothelial carcinoma of the bladder within 60 days prior to registration; the carcinoma must be stage T1 high-grade, stage CIS, or stage Ta high-grade
* Patients with mixed urothelial carcinoma and a glandular and/or squamous component will be eligible for the trial, but the presence of other histologic variants, pure adenocarcinoma, or pure squamous cell carcinoma, or pure squamous carcinoma in situ will make a patient ineligible
* Patients must have had all visible tumor resected completely within 60 days prior to registration; CIS disease is not expected to be completely excised; all patients must have tumor tissue from the histologic diagnosis of recurrence available for central pathology review submission; failure to submit these materials will make the patient ineligible for this study
* Patients must have had cystoscopy confirming no visible papillary tumor within 21 days prior to registration; (CIS disease is not expected to have been completely excised); if the transurethral resection of bladder tumor (TURBT) or bladder biopsy falls within 21 days of registration it will fulfill this criterion
* Patients must have had urine cytology within 21 days prior to registration; cytology for patients with CIS component is not expected to be negative for malignant cells; if the cytology for male patients with only Ta/T1 disease in the absence of CIS is positive for malignant cells, patient must have had a biopsy of the prostatic urethra within the previous six months
* All patients with T1 urothelial carcinoma at study entry must undergo re-TURBT within 60 days prior to registration, and must have evidence of uninvolved muscularis propria in the pathologic specimen from either the first or the second TURBT; tissue from the re-resection must be submitted for central review in addition to the tissue from the first TURBT; the TURBT that identified the recurrent T1 disease may have taken place more than 60 days prior to registration but not more than 120 days; patients with high grade Ta or CIS do not require a re-TURBT, but if this is performed at the discretion of the treating physician, the second TURBT must be within 60 days of registration; there is no requirement for muscularis propria in the specimen of Ta/CIS patients, but the tissue from the first and second TURBTs must be submitted for central review; if a patient with Ta/T1 disease undergoes repeat TURBT, the patient will be stratified as having CIS if there is CIS on either TURBT
* Patients must not have had urothelial carcinoma in the prostatic urethra within the previous 24 months or muscle invasive urothelial carcinoma of the bladder at any time; patients with prior urothelial carcinoma in the upper urinary tract within the previous 24 months will only be eligible if they had =< T1 carcinoma and were treated with nephroureterectomy; patients must have a computed tomography (CT) or magnetic resonance imaging (MRI) (including CT-intravenous pyelogram [IVP], CT-urogram or MR-urogram) of the abdomen and pelvis to rule out upper tract malignancy and intra-abdominal metastases within 90 days prior to registration; if a patient cannot tolerate intravenous contrast, a retrograde pyelogram should be performed within 90 days prior to registration
* Patients must be deemed unfit for radical cystectomy by the treating physician, or the patient must refuse radical cystectomy, which is considered standard of care for these patients; the reason for patients not to undergo cystectomy will be clearly documented
* Patients must be BCG-unresponsive; a patient is BCG-unresponsive if they meet one or more of the following criteria:

  * Patient has persistent or recurrent high-grade Ta/CIS urothelial carcinoma after completing therapy with at least induction BCG (>= 5 doses) and first round maintenance (>= 2 doses) or second induction BCG (>= 2 doses); both rounds of BCG must have been administered within a 12 month period; these patients must have either had high-grade Ta tumors and did not achieve a disease-free state for more than 6 months following last dose of BCG, or they had CIS and did not achieve a CR; S1605 registration must occur within 9 months of the last dose of BCG

    * If a patient does not meet these criteria only because the last dose of BCG was more than 9 months ago, the patient may become eligible if he/she shows histologically proven high-grade recurrence after an additional round of induction or maintenance BCG (>= 3 doses) within 9 months prior to registration
  * Patient has persistent or recurrent high grade T1 urothelial carcinoma after completing therapy with at least induction BCG (>= 5 doses); patients with recurrent high grade T1 urothelial carcinoma after additional rounds of BCG will also be eligible, but one round of maintenance therapy or a second induction is not a pre-requisite for these patients. Trial registration must occur within 9 months of the last dose of BCG

    * If a patient does not meet these criteria only because the last dose of BCG was more than 9 months ago, the patient may become eligible if he/she shows histologically proven high grade recurrence after an additional round of induction or maintenance BCG (>= 3 doses) within 9 months prior to registration
  * Patient achieves disease-free state at 6 month time point (i.e., complete response; presence of only low-grade tumor at this timepoint is still considered complete response) after induction and maintenance (or second round of induction) BCG but later experiences a high-grade Ta/T1 recurrence (with or without concomitant CIS) within 6 months after the last dose of BCG or recurrent CIS (in absence of concomitant Ta/T1 tumor) within 12 months after the last BCG dose; the time of eligibility is measured from the last dose of BCG to the time of disease recurrence; the patient must be registered on the trial within 60 days of this recurrence, or within 60 days of a re-TURBT if indicated
* All adverse events associated with any prior surgery and intravesical therapy must have resolved to grade =< 2 prior to registration
* Absolute neutrophil count (ANC) >= 1,500 microliter (mcL) (within 42 days prior to registration)
* Platelets >= 100,000/mcL (within 42 days prior to registration)
* Hemoglobin >= 9 g/dL (within 42 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL) (within 42 days prior to registration)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2 x IULN (within 42 days prior to registration)
* Serum creatinine =< 1.5 ULN OR measured or calculated creatinine clearance >= 30 mL/min (within 42 days prior to registration)
* Patients must have Zubrod performance status =< 2
* Patients must have a baseline electrocardiograph (ECG) performed within 42 days prior to registration
* Patients positive for human immunodeficiency virus (HIV) are eligible only if they have all of the following:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests
* No other prior malignancy is allowed except, for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must be offered the opportunity to participate in specimen banking for future studies, to include translational medicine studies
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the oncology patient enrollment network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Patients must not have had prior systemic chemotherapy for bladder cancer or systemic immunotherapy, including, but not limited to interferon alfa-2b, high dose interleukin 2 (IL-2), pegylated interferon (PEG-IFN), PD-1, anti-PD-L1, intra-tumoral; patients must not have had vaccine therapies within 6 weeks prior to registration; patients must not have received or be planning to receive any of the prohibited therapies during protocol treatment; prior intravesical administration of chemotherapy, interferon, Vicinium (VB4-485), BC-819 or Instiladrin (rAd-interferon-alpha/Syn3) is allowed if all other criteria are met and the last administration was >= 30 days before registration
* Patients must not be planning to receive concomitant other biologic therapy, radiation therapy, intravesical chemotherapy, surgery, or other anti-cancer therapy while on this protocol
* Patients must not have received any prior radiation to the bladder for bladder cancer
* Patients must not have received treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 4 weeks prior to registration; exceptions: (1) patients may have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea); (2) the use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients must not have received a live, attenuated vaccine within 4 weeks before registration or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Patients must not require treatment with a RANKL inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab
* Patient must not have history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis
* Patients must not have an active infection requiring oral or IV antibiotics within 14 days prior to registration; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Patients must not have severe infections within 28 days prior to registration, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Patients must not have active autoimmune disease that has required systemic treatment in past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; autoimmune diseases include, but are not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* Patients must not have undergone prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patient must not have active tuberculosis
* Patients must not have active hepatitis B (chronic or acute) or active hepatitis C infection

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* Patients must not be pregnant or nursing due to the potential teratogenic side effects of the protocol treatment; administration of atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Due to the potential drug reaction with atezolizumab, patients must not be known to be allergic to Chinese hamster egg or ovaries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Black, Principal Investigator — SWOG Cancer Research Network
Locations (272):
- United States (269):
  - Southern Cancer Center PC-Daphne, Daphne, Alabama
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale University, New Haven, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Reid Health, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai West, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - WG Hefner VA Medical Center, Salisbury, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Black PC, Tangen CM, Singh P, McConkey DJ, Lucia MS, Lowrance WT, Koshkin VS, Stratton KL, Bivalacqua TJ, Kassouf W, Porten SP, Bangs R, Plets M, Thompson IM Jr, Lerner SP. Phase 2 Trial of Atezolizumab in Bacillus Calmette-Guerin-unresponsive High-risk Non-muscle-invasive Bladder Cancer: SWOG S1605. Eur Urol. 2023 Dec;84(6):536-544. doi: 10.1016/j.eururo.2023.08.004. Epub 2023 Aug 16. PMID 37596191

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 172 participants were registered for the study: 101 on the CIS +/ Ta/T1 stratification and 71 on the Ta/T1 (without CIS) stratification. Six participants did not receive protocol therapy, leaving 166 participants were included in the safety analysis population: 96 on the CIS +/ Ta/T1 stratification and 70 on the Ta/T1 (without CIS) stratification. 37 participants were ineligible, leaving 129 eligible and evaluable total participants.
Groups:
- Atezolizumab - CIS +/ Ta/T1: Patients with CIS +/ Ta/T1 histology at baseline. Patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles (51 weeks) in the absence of disease progression or unacceptable toxicity.
  Atezolizumab: Given IV
- Atezolizumab - Ta/T1 (Without CIS): Patients with Ta/T1 (without CIS) histology at baseline. Patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles (51 weeks) in the absence of disease progression or unacceptable toxicity.
  Atezolizumab: Given IV
Period: Overall Study
Arm/Group | Atezolizumab - CIS +/ Ta/T1 | Atezolizumab - Ta/T1 (Without CIS)
Started | 101 | 71
Safety Analysis Population | 96 | 70
Eligible and Evaluable | 74 | 55
Completed | 13 | 20
Not Completed | 88 | 51
Not completed — No protocol treatment received | 5 | 1
Not completed — Ineligible | 22 | 15
Not completed — Participant refusal | 5 | 5
Not completed — Adverse Event | 5 | 4
Not completed — Death | 0 | 1
Not completed — Disease progression/recurrence | 50 | 24
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes the 129 participants that received protocol therapy and were eligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab - CIS +/ Ta/T1 | Atezolizumab - Ta/T1 (Without CIS) | Total
Number analyzed (Participants) | 74 | 55 | 129
Age, Continuous [Median (Full Range); unit: years] | 73 [47 to 90] | 74 [38 to 97] | 74 [38 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 62 | 46 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 70 | 49 | 119
  Other, unknown | 4 | 6 | 10
Zubrod Performance Status Score [Count of Participants; unit: Participants] — Zubrod performance status scores range from 0 to 5, with higher scores reflecting greater disability. Only participants with scores from 0 to 2 were eligible for this study.
  Participants
    0 | 57 | 36 | 93
    1 | 17 | 17 | 34
    2 | 0 | 2 | 2
Histology [Count of Participants; unit: Participants]
  CIS only | 43 | 0 | 43
  CIS + Ta | 14 | 0 | 14
  CIS + T1 | 13 | 0 | 13
  CIS + Ta + T1 | 4 | 0 | 4
  Ta only | 0 | 30 | 30
  T1 only | 0 | 22 | 22
  Ta + T1 | 0 | 3 | 3
Median Prior BCG Installations [Median (Full Range); unit: BCG instillations] — Bacillus Calmette-Guerin (BCG) is the main intravesical immunotherapy for early-stage bladder cancer.
  BCG instillations | 12 [6 to 29] | 12 [6 to 31] | 12 [6 to 31]
Median Time Since Last BCG [Median (Full Range); unit: Days] | 154 [5 to 346] | 127 [67 to 273] | 136 [5 to 346]
Reason for not Undergoing Cystectomy [Count of Participants; unit: Participants]
  Ineligible | 5 | 7 | 12
  Patient choice | 69 | 48 | 117

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate in the Subset of Patients With Carcinoma in Situ (CIS)
Description: To estimate complete response at 25 weeks after registration for those with a CIS component. Complete Response (CR) is defined as negative biopsy for high grade disease at Week 25 (± 7 days) for the subset of patients with a CIS component at study entry, according to local pathology call. In addition, patients with a CIS component who undergo negative biopsy at Week 13 for suspicious cystoscopy and or positive cytology and have cystoscopy not suspicious for cancer and cytology not positive for malignant cells at Week 25 do not require repeat biopsy at Week 25 and will be considered to have a complete response at Week 13 and will also be counted as having a complete response at Week 25.
Time Frame: At 25 weeks
Population: The analysis population included the 74 participants that had CIS +/ Ta/T1 histology, received protocol therapy, and were eligible for the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab - CIS +/ Ta/T1
Number analyzed (Participants) | 74
percentage of participants | 27 [17 to 38]

2. Primary Outcome: Event-free Survival (EFS)
Description: To evaluate event-free survival at 18 months in patients with BCG-unresponsive high-risk non-muscle invasive bladder cancer (Ta/T1/CIS) treated with atezolizumab. Event-Free Survival is defined as time from date of registration to first documentation of event. Participants last known to be alive and not to have recurred are censored at the date of last contact. An event was defined as the first occurrence of any of the following: biopsy-proven high-grade bladder cancer (including persistent CIS at 3 and/or 6 months); high-grade upper tract urothelial carcinoma; high-grade urothelial carcinoma of the prostatic urethra; muscle-invasive disease; clinical evidence of metastatic disease; or death due to any cause.
Time Frame: 18 months
Population: The two primary outcomes were hierarchical co-primary endpoints - CR rate in the CIS subset and 18-month EFS for all patients. The protocol states that EFS in all patients would only be evaluated if the CR rate in evaluable patients in the CIS subset was statistically significant. Because the primary endpoint of CR at 6 months for CIS patients did not meet pre-specified criteria, we did not conduct the analysis of EFS in all patients so there are no results to report for this endpoint.
Groups:
- Atezolizumab: Patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles (51 weeks) in the absence of disease progression or unacceptable toxicity.
Arm/Group | Atezolizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Event-free Survival (EFS) in the Ta/T1 Subset
Description: To evaluate event-free survival at 18 months in the subset of participants with papillary cancer (Ta/T1) treated with atezolizumab. Event-Free Survival is defined as time from date of registration to first documentation of event. Participants last known to be alive and not to have recurred are censored at the date of last contact. An event was defined as the first occurrence of any of the following: biopsy-proven high-grade bladder cancer (including persistent CIS at 3 and/or 6 months); high-grade upper tract urothelial carcinoma; high-grade urothelial carcinoma of the prostatic urethra; muscle-invasive disease; clinical evidence of metastatic disease; or death due to any cause.
Time Frame: 18 months
Population: Only participants who were eligible and received at least one dose or protocol therapy were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab - Ta/T1 (Without CIS)
Number analyzed (Participants) | 55
percentage of participants | 49 [34 to 57]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: To evaluate progression-free survival at 18 months in all eligible and evaluable participants. Progression-free survival (PFS) is defined as the time from registration to first evidence of biopsy-proven muscle-invasive bladder cancer (T>=2), nodal or distant metastasis, or death from any cause. Participants without an event were censored at the date of their last cystoscopy. Estimated using Kaplan-Meier.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 129
percentage of participants | 82 [74 to 88]

5. Secondary Outcome: Time to Cystectomy
Description: Time to cystectomy is defined as time from discontinuation of protocol therapy to time of cystectomy.
Time Frame: Up to 5 years
Population: This study is a single arm study and while other outcome measures compared the two strata (CIS +/ Ta/T1 and Ta/T1 (Without CIS)), the population for this outcome measure is unstratified and includes all 33 participants across both strata that underwent a radical cystectomy.
Measure: Median (Full Range); unit: days
Arm/Group | Atezolizumab
Number analyzed (Participants) | 33
days | 106 [33 to 1233]

6. Secondary Outcome: Bladder Cancer-Specific Survival
Description: To evaluate bladder cancer-specific survival at 3 years in all eligible and evaluable participants. Bladder cancer-specific survival is defined as the time from registration to death due to bladder cancer. Participants without bladder cancer death are censored at last contact date or date of non-bladder cancer death. Estimated using Kaplan-Meier.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 129
percentage of participants | 91 [83 to 95]

7. Secondary Outcome: Three-Year Overall Survival
Description: Overall survival (OS) is defined as the time from registration to the date of death due to any cause. Participants last known to be alive are censored at the date of last contact.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Atezolizumab - CIS +/ Ta/T1 | Atezolizumab - Ta/T1 (Without CIS)
Number analyzed (Participants) | 74 | 55
percentage of paticipants | 80 [70 to 90] | 79 [68 to 91]

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 5 years after registration
Description: Adverse events (AEs) are reported by CTCAE Version 4.0. 166 participants received at least one dose of protocol treatment and were assessed for adverse events and all-cause mortality
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 25/166
Serious Adverse Events (participants affected / at risk) | 42/166
Other Adverse Events (participants affected / at risk) | 161/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (N=166)
Anemia (Blood and lymphatic system disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Endocrine disorders-Other (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Device related infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations-Other (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
CPK increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Lipase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Nervous system disorders-Other (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 6
Renal and urinary disorders-Other (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures-Other (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab (N=166)
Anemia (Blood and lymphatic system disorders) | 39
Hyperthyroidism (Endocrine disorders) | 10
Hypothyroidism (Endocrine disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 24
Diarrhea (Gastrointestinal disorders) | 45
Nausea (Gastrointestinal disorders) | 23
Chills (General disorders) | 11
Edema limbs (General disorders) | 13
Fatigue (General disorders) | 84
Fever (General disorders) | 15
Flu like symptoms (General disorders) | 9
General disorders and admin site conditions - Other (General disorders) | 12
Pain (General disorders) | 15
Upper respiratory infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 20
Bruising (Injury, poisoning and procedural complications) | 9
Fall (Injury, poisoning and procedural complications) | 10
Alanine aminotransferase increased (Investigations) | 24
Alkaline phosphatase increased (Investigations) | 20
Aspartate aminotransferase increased (Investigations) | 31
Blood bilirubin increased (Investigations) | 11
Creatinine increased (Investigations) | 29
Investigations-Other (Investigations) | 12
Lymphocyte count decreased (Investigations) | 19
Platelet count decreased (Investigations) | 14
White blood cell decreased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 20
Hypercalcemia (Metabolism and nutrition disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 37
Hyperkalemia (Metabolism and nutrition disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 22
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 24
Insomnia (Psychiatric disorders) | 10
Hematuria (Renal and urinary disorders) | 20
Renal and urinary disorders-Other (Renal and urinary disorders) | 11
Urinary frequency (Renal and urinary disorders) | 15
Urinary tract pain (Renal and urinary disorders) | 10
Urinary urgency (Renal and urinary disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 33
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 27
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 24
Hypertension (Vascular disorders) | 28

LIMITATIONS AND CAVEATS:
There were two hierarchical co-primary endpoints, the analysis of the latter, event-free survival (EFS), was not conducted because the first co-primary endpoint, complete response (CR) at 6 months for participants with CIS, did not meet the prespecified criteria to warrant analysis of EFS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT02844816/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT02844816/ICF_001.pdf